CLINICAL TRIAL: NCT02806999
Title: The Therapeutic Effects of Combination of Insulin With Berberine on the Patients With Stess Hyperlipemia:a Prospective, Double Blind, Randomized, Placebo-controlled, Single-center Clinical Trial
Brief Title: The Therapeutic Effects of Insulin and Berberine on Stress Hyperglycemia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HYYuan; 20151025 (Other Grant/Funding Number: Traditional Chinese Medicine Bureau of Guangdong Province)
Record Dates: First submitted 2016-06-06; First posted 2016-06-21 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Hyperglycemia
Keywords: Heart disease; Postoperative period; Hyperglycemia; Berberine; Insulin; Clinical trials as topic
MeSH Terms: conditions — Hyperglycemia; Heart Diseases; Insulin Resistance | interventions — Berberine; Insulin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Berberine; Insulin (Experimental): Follow the previous administration program，participants will continue to receive intensive insulin therapy; Besides injecting insulin, participants will receive 500mg berberine twice a day for 8 days.
  Drug: Berberine; Insulin
  Interventions: Drug: Berberine; Insulin
- Insulin (Active Comparator): Besides receiving intensive insulin therapy, participants will take a placebo twice a day for 8 days.
  Drug: Insulin
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Berberine; Insulin — Participants will receive 500mg Berberine twice a day for 8 days; Meanwhile，participants will also continue to receive intensive insulin therapy.
  Other Names: No other name
  Arms: Berberine; Insulin
Drug: Insulin — Participants will continue to receive intensive insulin therapy; Meanwhile, Participants will also receive a placebo twice a day for 8 days.
  Other Names: No other name
  Arms: Insulin

SUMMARY:
Berberine is a conventional component in Chinese medicine. In recent years, effects of Berberine on improvement of glucose metabolism have been explored. The purpose of this study is to observe the therapeutic effects of combination of insulin and berberine on stress hyperglycemia in patients after cardiac surgery.

DETAILED DESCRIPTION:
Patients at risk for stress hyperglycemia are often prescribed insulin (Intensive insulin therapy, IIT and maintenance of blood glucose at a level between 80 and 110 mg per deciliter), which are the medication that reduce the level of glucose in the blood. By lowering the glucose level, these patients have a lower incidence of arrhythmia, myocardial ischemia and reperfusion injury, and heart failure and so on. But there are many patients whose hyperglycemia are not well controlled.If investigators are simply doubling the insulin, that only 10% of the benefit can be received.And it often bring significant side effects (Such as: hypoglycemia, etc.) in critically ill patients. Several studies have suggested that the use of berberine can effectively lowering the blood glucose level.The chemical structure and mechanisms of drug is clearly, and the side effects are seldom, the price of berberine is very cheap. The purpose of this study is to observe the therapeutic effects of combination of insulin and berberine on stress hyperglycemia in patients with heart disease whose level of blood glucose are not well controlled when only using insulin postoperatively.

This study will enroll postoperative patients who currently are injected with insulin by insulin pump，but the level of blood glucose is not controlled well. Patients will be assigned to receive 500mg of Berberine twice a day or a placebo(meanwhile they are receiving intensive insulin therapy) in a randomized, double blind, and prospective way. Investigators will occur at preoperative baseline, operating time and postoperative days 2, 4 and 8. Blood will be collected for laboratory testing, and acute physiology and chronic health evaluationⅡ and therapeutic intervention scoring system-28 will assess patient's condition at baseline and days 2, 4 and 8. At days 2, 4 and 8, medication efficacy will be also assessed and tests of blood glucose will be performed. Insulin count will be used to assess effectiveness of Berberine treatment at days 2, 4 and 8. Meanwhile, medication side effects will be monitored and the incidence of hypoglycemia or stool frequency are rigorously recorded at days 2, 4 and 8.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of stress hyperglycemia (fasting glucose >6.9 mmol/L or random glucose >11.1 mmol/L without evidence of previous diabetes);
* Worsening glycemic control;
* Individuals who had cardiac surgery before recruitment;
* Those who voluntarily sign the consent form after being fully informed and understanding the purpose and procedures of the study, characters of the disease, effect of medications, methods of related examinations, and potential risk/benefits of the study;

Exclusion Criteria:

* Individuals with a history of diabetes;
* Individuals who are not able to cooperate;
* Female of childbearing potential;
* Severe liver or renal disease, or cancer history;
* Individuals who are involved in designing, planning or performing this clinical trial;
* Individuals with any condition that could be worsened by supplemental Berberine;
* Individuals with severe gastrointestinal disease;
* Individuals with infectious diseases;
* Current participation in another clinical trial;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-03 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Evidence of effects of insulin and berberine on stress hyperglycemia | Within the first 10 days (plus or minus 3 days) after cardiac surgery
  Levels of blood glucose will be used to evaluate the hypoglycemic activity of berberine (Blood glucose is measured every 4 hours, and when patient's blood glucose are not stable, blood glucose can be measured every 1 hours.).

SECONDARY OUTCOMES:
Synergy of insulin and berberine on stress hyperglycemia | Within the first 10 days (plus or minus 3 days) after cardiac surgery
  Total dose of insulin (If there is synergy between insulin and berberine, the total dose of insulin should be reduced.)
Mechanism of berberine on stress hyperglycemia | Within the first 10 days (plus or minus 3 days) after cardiac surgery
  Hyperinsulinaemic-euglycaemic clamp will be used to assess the improvement in insulin resistance and initially explore the mechanism of berberine hypoglycemic.

OTHER OUTCOMES:
Stool frequency | Within the first 10 days (plus or minus 3 days) after cardiac surgery
  Evaluating the side effects of Berberine (Causing constipation)
Incidence of hypoglycemia | Within the first 10 days (plus or minus 3 days) after cardiac surgery
  If the incidence of hypoglycemia is reduced, we will conclude that berberine can reduce the side effects of intensive insulin treatment.
Assessment of ventricular function by ultrasound | Within the first 10 days (plus or minus 3 days) after cardiac surgery
  EF (ejection fraction) value will be measured by ultrasound to assess cardiac function.
Intensive care time | Within the first 10 days (plus or minus 3 days) after cardiac surgery
All cause mortality | Within the first 10 days (plus or minus 3 days) after cardiac surgery
Assess the severity of the disease by APACHEⅡ | Within the first 10 days (plus or minus 3 days) after cardiac surgery
  The full name of APACHEⅡ is acute physiology and chronic health Ⅱ, a questionnaire is used to acess the severity of the disease.
Assess the nursing workload by TISS-28 | Within the first 10 days (plus or minus 3 days) after cardiac surgery
  The full name of TISS-28 is therapeutic intervention scoring system-28. It is a questionnaire used to assess the nursing workload in ICU patients, so TISS-28 can indirectly reflect patient's condition.
Incidence of nosocomial infections | Within the first 10 days (plus or minus 3 days) after cardiac surgery
  Stress hyperglycemia leads to decreased immunity, and good blood glucose control helps to reduce nosocomial infections.

CONTACTS AND LOCATIONS:
Overall Officials: Weiping Xiong, M.D., Principal Investigator — Guangdong Cardiovascular Insititution, Guangdong General Hospital, Guangdong Academy of Medical Science
Locations (1):
- Guangdong Cardiovascular Insititution, Guangdong General Hospital, Guangdong Academy of Medical Science, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
Whether individual participant collected in this study data can be available depends on the participant's permission.

REFERENCES:
- [Background] Donnor T, Sarkar S. Insulin- Pharmacology, Therapeutic Regimens and Principles of Intensive Insulin Therapy. 2023 Feb 15. In: Feingold KR, Adler RA, Ahmed SF, Anawalt B, Blackman MR, Chrousos G, Corpas E, de Herder WW, Dhatariya K, Dungan K, Hamilton E, Hofland J, Jan de Beur S, Kalra S, Kaltsas G, Kapoor N, Kim M, Koch C, Kopp P, Korbonits M, Kovacs CS, Kuohung W, Laferrere B, Levy M, McGee EA, McLachlan R, Muzumdar R, Purnell J, Rey R, Sahay R, Shah AS, Sperling MA, Stratakis CA, Trence DL, Wilson DP, editors. Endotext [Internet]. South Dartmouth (MA): MDText.com, Inc.; 2000-. Available from http://www.ncbi.nlm.nih.gov/books/NBK278938/ PMID 25905175
- [Background] Dungan KM, Braithwaite SS, Preiser JC. Stress hyperglycaemia. Lancet. 2009 May 23;373(9677):1798-807. doi: 10.1016/S0140-6736(09)60553-5. PMID 19465235
- [Background] van den Berghe G, Wouters P, Weekers F, Verwaest C, Bruyninckx F, Schetz M, Vlasselaers D, Ferdinande P, Lauwers P, Bouillon R. Intensive insulin therapy in critically ill patients. N Engl J Med. 2001 Nov 8;345(19):1359-67. doi: 10.1056/NEJMoa011300. PMID 11794168
- [Background] Rassias AJ. Intraoperative management of hyperglycemia in the cardiac surgical patient. Semin Thorac Cardiovasc Surg. 2006 Winter;18(4):330-8. doi: 10.1053/j.semtcvs.2006.05.002. PMID 17395030
- [Background] Lee YS, Kim WS, Kim KH, Yoon MJ, Cho HJ, Shen Y, Ye JM, Lee CH, Oh WK, Kim CT, Hohnen-Behrens C, Gosby A, Kraegen EW, James DE, Kim JB. Berberine, a natural plant product, activates AMP-activated protein kinase with beneficial metabolic effects in diabetic and insulin-resistant states. Diabetes. 2006 Aug;55(8):2256-64. doi: 10.2337/db06-0006. PMID 16873688
- [Background] Wiener RS, Wiener DC, Larson RJ. Benefits and risks of tight glucose control in critically ill adults: a meta-analysis. JAMA. 2008 Aug 27;300(8):933-44. doi: 10.1001/jama.300.8.933. PMID 18728267
- [Background] Monzillo LU, Hamdy O. Evaluation of insulin sensitivity in clinical practice and in research settings. Nutr Rev. 2003 Dec;61(12):397-412. doi: 10.1301/nr.2003.dec.397-412. PMID 14968910
- [Background] Capes SE, Hunt D, Malmberg K, Gerstein HC. Stress hyperglycaemia and increased risk of death after myocardial infarction in patients with and without diabetes: a systematic overview. Lancet. 2000 Mar 4;355(9206):773-8. doi: 10.1016/S0140-6736(99)08415-9. PMID 10711923
- [Background] Geng FH, Li GH, Zhang X, Zhang P, Dong MQ, Zhao ZJ, Zhang Y, Dong L, Gao F. Berberine improves mesenteric artery insulin sensitivity through up-regulating insulin receptor-mediated signalling in diabetic rats. Br J Pharmacol. 2016 May;173(10):1569-79. doi: 10.1111/bph.13466. Epub 2016 Apr 5. PMID 26914282
- [Background] Zhao GL, Yu LM, Gao WL, Duan WX, Jiang B, Liu XD, Zhang B, Liu ZH, Zhai ME, Jin ZX, Yu SQ, Wang Y. Berberine protects rat heart from ischemia/reperfusion injury via activating JAK2/STAT3 signaling and attenuating endoplasmic reticulum stress. Acta Pharmacol Sin. 2016 Mar;37(3):354-67. doi: 10.1038/aps.2015.136. Epub 2016 Jan 25. PMID 26806299
- [Background] Agus MS, Asaro LA, Steil GM, Alexander JL, Silverman M, Wypij D, Gaies MG; SPECS Investigators. Tight glycemic control after pediatric cardiac surgery in high-risk patient populations: a secondary analysis of the safe pediatric euglycemia after cardiac surgery trial. Circulation. 2014 Jun 3;129(22):2297-304. doi: 10.1161/CIRCULATIONAHA.113.008124. Epub 2014 Mar 26. PMID 24671945
- See also: Click here for more information about this study: Therapeutic Effects of Berberine in Patients With Type 2 Diabetes — https://clinicaltrials.gov/ct2/show/record/NCT00425009?term=berberine&rank=13